Ase I, Randomized, Open-label, Single-dose, 2-way Crossov ady to Compare the Pharmacokinetics of Budeson Delivere by PT027 to Pulmicort Respules® in Children with Asthma Aged 4 to 8 Years (BLANC) A Phase I, Randomized, Open-label, Single-dose, 2-ways Crossover Study to Compare the Pharmacokinetics of Budeson de Delivered by PT027 to Pulmicort Respules® in Children with Asthmatical to 8 Years (BLANC) A Phase I, Randomized, Open-label, Single-dose, 2-ways Crossover Study to Compare the Pharmacokinetics of Budeson de Delivered by PT027 to Pulmicort Respules® in Children with Asthmatical Asthmatical Compared to 8 Years (BLANC)

Study Statistician

This document must not be used to support any marketing.

A Phase I, Randomized, Open-label, Single-dose, 2-way Crossover application Study to Compare the Pharmacokinetics of Budesonide Delivered by PT027 to Pulmicort Respules® in Children to 8 Years (RI ANG) by PT027 to Pulmicort Respules® in Children with Asthma Aged 4 to 8 Years (BLANC)

Avillion Statistician

This document must not be used to support any marketing at most decimal transfer of the standard of the standa

# Contents

| 1. | STUDY DETAILS | 8 |
|---|---|---|
| 1.1 | Study objectives | 8 |
| 1.1.1 | Primary objective | |
| 112 | Secondary objective | |
| 113 | Safety objective | |
| | Exploratory objective | 8 |
| 1.1.7 | Ct. 1. 1. i | |
| 1.2 | Study design | |
| 1.3 | Number of subjects | ç¥1 |
| 1.3.1 | Randomization | GS11 |
| 1.3.2 | Sample Size Calculation | 211 |
| 2. | ANALYSIS SETS AND PROTOCOL DEVIATIONS | 11 |
| 2.1 | Definition of analysis sets | 11 |
| 2.1.1 | Pharmacokinetic (PK) analysis set | 11 |
| 2.1.2 | Safety analysis set | 11 |
| 2.1.3 | All subjects enrolled analysis set | 12 |
| 2.1.4 | All subjects randomized analysis set | 12 |
| 2.2 | Protocol deviations | 12 |
| 3. | Exploratory objective Study design Number of subjects Randomization Sample Size Calculation ANALYSIS SETS AND PROTOCOL DEVIATIONS Definition of analysis sets Pharmacokinetic (PK) analysis set Safety analysis set All subjects enrolled analysis set All subjects randomized analysis set Protocol deviations PRIMARY AND SECONDARY VARIABLES General Definitions Screening period Crossover periods Derivation of PK parameters Primary endpoints Primary endpoints Secondary endpoints Safety variables Safety variables Safety variables | 12 |
| 3.1 | General Definitions | 12 |
| 3 1 1 | Screening period | 12 |
| 3.1.2 | Crossover periods | 13 |
| 3.1.3 | Derivation of PK parameters 2 | 13 |
| 3.1.4 | Relative time from first dose of randomized treatment | 13 |
| 3.1.5 | Visit windowing | 14 |
| 3.1.6 | Imputation rules | 14 |
| 3.2 | Primary endpoints | 16 |
| 3.3 | Secondary endpoints | 16 |
| 3.4 | Safety variables | 16 |
| 3.4.1 | Vital signs | 16 |
| 3.4.2 | Adverse Events (including Serious Adverse Events) | 17 |
| 3.4.3 | Laborstory Safety Variables | 19 |
| 3.5 | Qtber variables | 20 |
| 3.5.1 | Prior and Concomitant medications | 20 |
| 3.5.2 <b>3</b> | Withdrawal from study | 20 |
| 3.5.3 | Screen Failures | 21 |
| ther. | Vital signs Adverse events (including Serious Adverse Events) Laboratory Safety Variables Other variables Prior and Concomitant medications Withdrawal from study Screen Failures ANALYSIS METHODS Statistical Considerations | 22 |
| 4.1 | Statistical Considerations | 22 |
| 4.1.1 | Treatment groups | 22 |
| 4.2 | Analysis methods | 22 |
| 4.2.1 | Subject Disposition | |
| 4.2.2 | Demographic and Baseline Characteristics. | 23 |

| | Statistical A<br>AV006 1.0 | nalysis Plan | Avillion |
|---|---|---|---|
| | 4.2.3<br>4.2.4<br>4.2.5<br>4.2.6<br>4.2.7 | Treatment Exposure Protocol deviations Pharmacokinetics (PK) Analysis of safety variables COVID-19 impacts | 24<br>24<br>25<br>27<br>29 |
| | 5. | CHANGES OF ANALYSIS FROM PROTOCOL | 30 application |
| | | Treatment Exposure Protocol deviations. Pharmacokinetics (PK) Analysis of safety variables COVID-19 impacts CHANGES OF ANALYSIS FROM PROTOCOL. CHANGES OF ANALYSIS FROM PROTOCOL. CHANGES OF ANALYSIS FROM PROTOCOL. CHANGES OF ANALYSIS FROM PROTOCOL. Analysis of safety variables COVID-19 impacts CHANGES OF ANALYSIS FROM PROTOCOL. | |
| This doc | Junent must | Lingt D. | |

CONFIDENTIAL AND PROPRIETARY

# LIST OF FIGURES

| LIST OF FIGURES | S | |
|---|---|---|
| Figure 1: Study schema. | 9 | ation |
| LIST OF TABLES | ents and procedures | applica |
| Table 1: Study assessme | ents and procedures | ۶ |
| Table 2: Laboratory Safe | ety Variables | |
| Table 2. Laboratory Sar | ASION 1 | |
| | ter. | |
| LIST OF ABBREV | TATIONS | |
| LIST OF HUDDREY | non non | |
| Abbreviation or special | Explanation | |
| term | Explanation | |
| AE | Adverse event | |
| ANOVA | Analysis of variance | |
| AUC0-inf | Area under the plasma concentration-time cove from time zero to infinity | |
| AUC0-t | Area under the plasma concentration-time curve from time zero to immity Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration Budesonide/albuterol sulfate Budesonide/albuterol sulfate Body mass index Drug concentration at law observed (quantifiable) concentration Maximum observed flasma concentration Case report form Clinical study protocol | |
| 11000 | quantifiable concentration | |
| BDA | Budesonide/albuterol sulfate | |
| BDA MDI (PT027) | Budesonide/albuterol sprice pered-dose inhaler | |
| BMI | Body mass index | |
| Clast | Drug concentration at last observed (quantifiable) concentration | |
| Cmax | Maximum observed plasma concentration | |
| CRF | Case report form | |
| CSP | Clinical study protocol | |
| eCRF | Electronic ase report form | |
| IMP | Investigational medicinal product | |
| λz | Terminal elimination rate constant | |
| LAR | Regally authorized representative | |
| MDI | Metered-dose inhaler | |
| MDI MedDRA NCA | Medical Dictionary for Regulatory Activities | |
| NCA US | Non-compartmental analysis | |
| PK V | Pharmacokinetic(s) | |
| PT , CO | Preferred term | |
| SAE NS | Serious adverse event | |
| sog | System Organ Class | |
| TAR | Treatment-emergent adverse event | |
| PK PT SAE SORTHUS TRAE | Half-life associated with terminal slope (λz) of a semi-logarithmic | |
| 1/2/12 | concentration-time curve | |
| tlast | Time of last quantifiable plasma concentration | |
| tmax | Time to reach maximum observed plasma concentration | |
| TC | Telephone call | |

# AMENDMENT HISTORY

| Date | Brief description of change |
|------|-----------------------------|
| | N/A |

The statement and the seed to separate any national and the seed to see a seed to seed to see a seed to see a seed to see a seed to see a seed to seed to see a seed to see a seed to see a seed to see a seed to seed to see a seed to see a seed to see a seed to see a seed to seed to see a

#### 1. STUDY DETAILS

#### Study objectives 1.1

#### Primary objective 1.1.1

| Primary Objective: | Primary endpoint: |
|---|---|
| To determine and compare the systemic exposure of budesonide after single-dose administrations of BDA MDI and Pulmicort Respules. | AUC0-t and Cmax |
| 1.1.2 Secondary objective | d oxig. |
| 0 1 011 1 | |

#### 1.1.2 Secondary objective

| Secondary Objective: | Secondary endpoint: |
|---|---|
| To determine and compare other PK<br>parameters for budesonide delivered by<br>BDA MDI and Pulmicort Respules | tmax, tlast, t½λz, λz, Clast and AUC0-inf (if feasible) |

#### 1.1.3 Safety objective

| Safety objective: | Safet Sendovints: |
|------------------------------------------|-------------------|
| To assess the safety and tolerability of | AGS/SAES |
| BDA MDI and Pulmicort Respules | CKC alle |

AE: adverse event; AUC0-inf: area under the plasma concentration-time curve from time zero to infinity; AUC0-t: area under the plasma concentration-time curve from time zero to time of last quantifiable concentration; BDA MDI: budesonide/albuterol sulfate metered-dose inhafer; Clast: drug concentration at last observed (quantifiable) timepoint; Cmax: maximum observed plasma comentration; PK: pharmacokinetic; SAE: serious adverse event. tlast: time of last quantifiable plasma concentration; tmax: time to reach maximum observed plasma concentration; t½λz: half-life associated with terminal slow (λz) of a semi-logarithmic concentration-time curve.

# Exploratory objective

Exploratory objectives are por planned for this study.

### Study design 1.2

This is a randomised, multicenter, open-label, single-dose, 2-way crossover study to compare the systemic exposure of budesonide delivered by the combination inhaler (BDA MDI 160/180 ug) with Pulmicort Respules 1 mg. The study consists of a screening visit (Visit 1) and 2 treatment visits (Wisit 2 and Visit 3). Randomization takes place at Visit 2. A follow-up (or early

with a wal, if applicable) telephone call (TC) will occur 2 to 5 days after the last dose.

See Figure 1 for a graphical presentation of the study design and Table 1 for a list of study assessments, as per protocol.

Figure 1: Study schema



Table 1: Study assessments and procedures

| | Screening<br>Period | | el Treatment<br>eriod | Follow-up or earl<br>withdrawal |
|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 - TC |
| Day | Starting from<br>Day -14 | 1 | 2 to 14 days<br>after V2 | 2 to 5 days after<br>V3 |
| Informed consent/assent | X | | | |
| Eligibility criteria | X | | | |
| Re-check eligibility criteria | | X | | 48 |
| Randomization | | X | | :00 |
| Routine clinical procedures | | | | Leinste |
| Medical/surgical history | X | | | ete |
| Demography | X | | | 70, |
| Physical examination | X | | | <u> </u> |
| Height, weight, and BMI | X | | Yall | |
| Routine safety measurements | | | KING | |
| Laboratory assessments (including<br>local laboratory clinical chemistry,<br>hematology, and urinalysis) a | X | الم الم | ionor | |
| AEs and concomitant medications | X | OR YOU | X | X |
| Seated vital signs (blood pressure<br>and heart rate) b | X AD | ation X | х | |
| Placebo MDI training c | W voll | | | |
| Nebulization training | QEX guit | | | |
| Randomized IMP | Ping | X | X | |
| Informed consent/assent Eligibility criteria Re-check eligibility criteria Randomization Routine clinical procedures Medical/surgical history Demography Physical examination Height, weight, and BMI Routine safety measurements Laboratory assessments (including local laboratory clinical chemistry, hematology, and urinalysis) a AEs and concomitant medications Seated vital signs (blood pressure and heart rate) b Placebo MDI training c Nebulization training Randomized IMP Blood sampling for PK - Timepaints AE: adverse event; By body mass index. min: minute; PK: planmacokinetic; TC: tel a Laboratory assessments (clinical chemist Study Protocol (CSP), Section 6.3.1. | Raite | A total o<br>will be<br>treatm<br>pre-dose<br>40, 60, 1<br>480, and | of 10 samples<br>taken per<br>ent visit at<br>and at 10, 20,<br>20, 240, 360,<br>720 min after<br>osing. | |
| AE: adverse event; Blee. body mass index. min: minute; PK: platmacokinetic; TC: tel a Laboratory assessments (clinical chemist Study Protocol (CSP), Section 6.3.1. b Vital signs will be assessed at the beginn c Training for placebo MDI will occur at V training prior to randomization. | mig (pre-dose) and | the end (post | -last PK sample) | of each study visit. |

# 1.3 Number of subjects

The target population will be male and female children with asthma, 4 to 8 years of age. Approximately 28 children will need to be screened, assuming an estimated screen failure rate of 50% prior to randomization in order for 14 children to be randomized and 10 to complete. At least 4 children should be randomized in the age range of 4-5 years. Children who do not complete both treatments (BDA MDI and Pulmicort Respules) may be replaced.

# 1.3.1 Randomization

At Visit 2, eligible subjects are randomized (1:1) to receive 1 of 2 treatment sequences BDA MDI 160/180 / Pulmicort Respules or Pulmicort Respules / BDA MDI 160/180). Randomization is stratified by study center, so that all subjects can be recruited at a single study center if needed.

# 1.3.2 Sample Size Calculation

No prospective calculations of statistical power have been made. At the study is descriptive with no formal hypothesis tests, complete data (evaluable data from both BDA MDI and Pulmicort Respules) from 10 children is considered sufficient to provide estimates of the PK parameters in this population without exposing more children than necessary to the IMP. Results will be interpreted in the perspective of the explorative nature of the study.

# 2. ANALYSIS SETS AND TO COL DEVIATIONS

# 2.1 Definition of analysis sets

# 2.1.1 Pharmacokinetic (PK) analysis set

The PK analysis set will consist of all randomized children for whom at least 1 of the primary PK parameters (AUC0-t and max) can be calculated and who have no important protocol deviations impacting the interpretation of the PK data.

Children who do not provide evaluable data for both treatments (BDA MDI and Pulmicort Respules) will be excluded from the analysis of variance (ANOVA).

Any excluded cases will be documented together with the reason for exclusion.

Profiles belonging to the PK analysis set will be summarized and analyzed according to the treatment that was administered at the specific visit. Any treatment errors will be documented as protocol deviations. All PK summaries will be based on the PK analysis set.

# 2.1.2 Safety analysis set

The safety analysis set is defined as all children receiving any amount of randomized treatment.

Occurrences of safety events (ie, AEs and use of concomitant medication) will be summarized under the actual treatment corresponding to the treatment period of which the event occurred. All safety summaries will be based on the safety analysis set.

and whose parent(s) or legally authorized representative(s) (LAR) have provided informed consent. This analysis set will be used for descriptive summaries of dispositions and subjects randomized analysis set.

All subjects randomized analysis set will be all or randomized to a treat.

The all subjects randomized analysis set will be defined as all children who have been randomized to a treatment sequence. This analysis set will be used to a suppose of the suppose of t randomized to a treatment sequence. This analysis set will be used for listing and descriptive summaries of demographic variables.

Subjects will be listed and summarized according to their randomized treatment sequence.

#### 2.2 Protocol deviations

A protocol deviation is any change, divergence, or departure from the study design or procedures defined in the protocol. Major protocoldeviations are defined as a subset of protocol deviations that may significantly affect the completeness, accuracy, and/or reliability of the study data or that may significantly affect subject's rights, safety, or well-being. Important protocol deviations (IPDs) are subset of major PDs deemed to impact the pharmacokinetics or the safety profit study. Minor PDs are the protocol deviations which are neither major nor important

Subjects must meet the eligibility criteria, assessed during screening, to be randomized to treatment. The list of inclusion and exclusion criteria are provided in the protocol. Eligibility criteria not met are collected on the electronic case report form (eCRF). Any children who do not fulfil all the eligibility criteria, but they are subsequently randomized in error and children who are erroneous prandomized will be identified as IPDs. Other IPDs may be identified by the sponsor prior the primary database lock.

A per protosol analysis excluding subjects with IPDs is not planned.

# PRIMARY AND SECONDARY VARIABLES

# General Definitions

# Screening period

Screening assessments are collected at Visit 1 (see Table 1). Any re-screening assessments that may occur (see 3.5.3) will be collected at Re-Screening visit.

#### 3.1.2 Crossover periods

Subjects will be randomized to a particular sequence and will receive the first treatment in their sequence at Visit 2 and second treatment at Visit 3. Period 1 corresponds to the results collected at Visit 2 and Period 2 corresponds to results collected at Visit 3. The below table represents planned treatment group assignment based on randomized sequence and crossover period.

| Randomized Treatment | Planned t | reatment group |
|---|---|---|
| Sequence | Period 1 (Visit 2) | Period 2 (Visit 3) |
| BDA MDI 160/180;<br>Pulmicort Respules | BDA MDI 160/180 | Pulmicort Resputes |
| Pulmicort Respules;<br>BDA MDI 160/180 | Pulmicort Respules | BDA 160/180 |

Pulmicort Respules is administered as a single dose of 1 mg.

3.1.3 Derivation of PK parameters

Plasma samples will be analyzed using non-comparing out analysis (NCA) to determine the Ost &, t½λz, and AUC0-inf [if feasible]) of PK parameters (AUC0-t, Clast, Cmax, tmax

budesonide in plasma.

A separate PK analysis plan, author by the PK specialists, will contain the derivation specifications of the PK parameters to delivered to

The derived PK parameters received from the PK specialists will be mapped to SDTM.PP, which will subsequently be propped to ADAM.ADPP. The latter analysis dataset will be used for programming data listories and descriptive summaries of the PK parameters.

#### Relative of the from first dose of randomized treatment 3.1.4

Plasma concentrations of budesonide will be measured in blood samples taken at planned timepoints (See Table 1). The actual timepoints with reference to the time of first dose of randomized treatment will be calculated separately for each visit (Visit 2 and Visit 3) as:

documents dose (hh:mm)]. [Relative time from first dose (minutes)] = [actual time of blood sample (hh:mm)] - [time of

Times of blood samples and time of first dose at the scheduled visits will be recorded on the eCRF at site.

#### 3.1.5 Visit windowing

Due to the design of this trial, there will be no visit windowing applied. Any unscheduled visits which may occur will not be used in analyses, however all data will be listed where

If a return to lockdown is announced or the study center is on lockdown and cannot process a visit, if possible, visits should be rescheduled to earlier/later as required to safeguard, salvient and study center staff.

3.1.6 Imputation rules

and study center staff.

3.1.6 Imputation rules

The following imputation rules will be applied to the raw data in order to calculate the PK and Safety analyses.

3.1.6.1 Missing date/time imputations

When determining whether concomitant medication or adverse event emergence is pre- or post-randomized treatment, the following imputation methods will be applied.

post-randomized treatment, the following imputation methods will be applied.

# Partial end date

- 1. If missing day [--/mm/yyyy] then simple as minimum (the end of the month, end of study participation).
- the impute as minimum {[31/12/yyyy], end of study 2. If missing month [--/ participation).
- 3. If completely missing, the set to end of study participation.

# Partial start date

- -/mm/yyyy] then impute as the minimum of:
- 1. If missing days Port and If mm/yyyy is the same as the dose date of BDA MDI then set to dose date of DA MDI; else if mm/yyyy is the same as the dose date of Pulmicort Respules then set to dose date of Pulmicort Respules; else set to 01/mm/yyyy
  - End date of medication/ event (after partial date handling has been applied).

missing month [--/--/yyyy] then impute as the minimum of:

- If yvvv same year as BDA MDI then set to date of BDA MDI dose; else if yyyy same year as Pulmicort Respules dose date set to dose date of Pulmicort Respules; Else set to start of the year [01/01/yyyy].
- End date of medication/ event (after partial date handling has been applied).
- If completely missing, then impute as the minimum of:

- Date of first dose of BDA MDI, unless missing then date of first dose of Pulmicort Respules.
- End date of medication/ event (after partial date handling has been applied).

profile, then they will be set as missing for the calculation of the descriptive summary statistics. Else if they occur prior to a quantifiable ......... statistics. Else if they occur prior to a quantifiable value, or no quantifiable value is provided within a visit-specific concentration profile, then they will be set to 0 for the calculation of the descriptive summary statistics. The original value will be listed.

#### Primary endpoints 3.2

The following PK parameters are of key interest for evaluating the systemic exposure of budesonide after single-dose administrations of BDA MDI and Pulmicort Respules.

3.3 Secondary endpoints
In addition to the above, the following parameters will be calculated to further askers the pharmacokinetics of BDA MDI compared to Pulmicort Respules:

• tmax: time to reach maximum observed plasma concentration
• tl/\(\lambda z\): half-life associated with terminal slope (\(\lambda z\)) and the semi-logarithmic concentration-time curve!

• \(\lambda z\): terminal elimination rate constant. It is additional to the semi-logarithmic concentration at the semi-lo

- AUC0-inf: area under the plastera concentration-time curve from time zero to infinity<sup>1</sup>

<sup>1</sup> Feasibility of endpoint provision will be determined by the PK specialist vendor.

# Safety variables 3.4

# Vital sign 3.4.1

The following vital signs measurements will be collected at screening Visit 1 and before dose and after the last blood sample is taken at Visit 2 and Visit 3 as per Table 1.

Qulse rate (beats/min)

Systolic blood pressure (mmHg)

Diastolic blood pressure (mmHg)

Any clinically significant changes in vital signs are recorded as an AE if applicable.

#### 3.4.2 Adverse events (including Serious Adverse Events)

#### 3.4.2.1 Definition of adverse event

An AE is the development of any untoward medical occurrence in a subject or clinical study to the medicinal product.

The term AE is used to include both serious and non-serious AEs and can include a sign deterioration of a pre-existing medical occurrence. An AE may occur at any time term and the screening period, even if no randomized treatment.

A treatment-emergent adverse event (TEAE) is defined as an AE with itset (start date/time) on or after the first dose of randomized IMP at Visit 2. Any AEs occurring in the washout between successive treatment periods will also be regarded as treatment-emergent and assigned to the treatment administered in the period prior to the washout.

3.4.2.2 Definition of serious adverse event

An SAE is an AE occurring during any study place. Fe., after the signing of the informed that fulfills 1 or more of the following consent/assent through to the safety follow Is immediately life-threatening eling author
Requires in-patient hospitalization. criteria:

- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or spirificant disability or incapacity
- Is a congenital abnormality or birth defect
- Is an important medical event that may jeopardize the subject or may require medical intervention prevent 1 of the outcomes listed above

All SAEs will be identified by the investigator and entered in the eCRF. The 'Serious?' field will be sento 'Y'.

Es and SAEs will be collected from time of signature of informed consent/assent, through the safety follow-up TC.

The following variables will be collected on the eCRF for each AE:

AE term (verbatim)

- Date/time when the AE started and stopped
  - DD/MMM/YYYY
- Maximum severity
- Seriousness
- Investigator causality rating against the randomized treatment
- Action taken with regard to the randomized treatment

  - Drug interrupted

  - Not applicable
- Outcome

  - Recovered/resolved with sequelae

  - Fata1

Anverse events data handling

Adverge events will be reported as starting during screening if the AE start date/time is prior

The first dose of randomized treatment taken at Visit 2.

Note that the first dose of randomized treatment at Visit 2.

Note that the first dose of randomized treatment at Visit 2. the first dose of randomized treatment at Visit 2. Any AEs occurring in the washout between successive treatment periods will also be regarded as treatment emergent and assigned to the actual treatment administered in the period prior to the washout.

andomized treatment

the randomized treatment

ed

areased

ose reduced

Drug interrupted

Drug permanently discontinued

Red attrotation applicable

ome

ecovered/resolved

covering/resolving manual red

covered/resolved

cover

If an AE has a missing onset date/time, then, unless the stop date/time of the AE indicates otherwise, this will be considered as treatment emergent. Similarly, if an AE has a partial onset date/time, then unless the partial onset date/time or the stop date/time indicates Please refer to Section 3.1.6 for the imputation rules to programmatically determine the of classification of AEs when there is partial start and/or stop dates recorded.

3.4.3 Laboratory Safety Variables

Samples for determination of clinical chemistry, hematology, and urinalysis will be taken at Visit 1 and at unscheduled visits, if required, as indicated in Table 2.

Additional safety samples may be collected if clinically indicated on the discontinuous formula to the disc otherwise, this will be considered as treatment emergent. AEs will be represented under the

Investigator.

The clinical chemistry, hematology, and urinalysis a session of the discretion of the d local laboratory. Sample tubes and sample sizes on a sample sizes of the sample sizes used and routine practice at each study center

Table 2: Laboratory Safety Variable

| Hematology/Hemostasis (whole blood) | Clinical Chemistry (serum or plasma) |
|---|---|
| Hematology/Hemostasis (whole blood) Basophils (%) Basophils Abs | Albumin |
| Basophils Abs | Alanine aminotransferase |
| Eosinophils (%) | Alkaline phosphatase |
| Eosinophils Abs | Aspartate aminotransferase |
| Hemoglobin SUP | Bilirubin, total |
| Eosinophils (%) Eosinophils Abs Hemoglobin Hematocrit Mean Corpus and Hemoglobin | Calcium, total |
| Mean Corpuscular richiogroum | Chloride |
| Mean Conguscular Hemoglobin Concentration | Cholesterol, total |
| Mean Corpuscular Volume | Creatinine |
| Mean corpuscular Volume | Creatine kinase |
| Monocytes Abs | Gamma-glutamyl transferase |
| Neutrophils (%) | Glucose (random) |
| Neutrophils Abs | Magnesium |
| Red blood cells (erythrocytes) | Phosphate |

| White blood cells (leukocytes) | Potassium |
|--------------------------------|-------------------|
| Platelet count | Protein, total |
| Lymphocytes Abs | Sodium |
| Lymphocytes (%) | Triglycerides |
| Urine* | |
| Urine blood | |
| Leukocyte esterase | - · |
| Urine protein | · or o |
| Urine glucose | or extension of s |
| Nitrite | |

Abs: absolute
\*If leukocyte esterase is detected, the site should send the sample for culture. If abnormal levels of blood or protein are detected, the sample should be sent for microscopic examination.

3.5 Other variables

3.5.1 Prior and Concomitant medications

The collection and recording of all concomitant medication, including all pre-enrollment asthmat therapies, are performed at each of the collection and recording of the collection. asthma therapies, are performed at each of the scheduled visits as detailed in Table 1.

All medications taken within 3 months before with 1 will be recorded as prior medications.

Any medication taken on or after Visit Daniel brough the follow-up TC will be recorded as concomitant therapy. All medications (prover and concomitant) will be recorded on the eCRF throughout the study.

Disallowed medications will be identified by a physician on review of the data which will be

completed prior to database ock. All identified medications which are disallowed will be considered for flagging and IPD during the protocol deviation reviews, prior to database lock.

If a concomitant medication is recorded with partial start date and/or end date of administration, a conservative approach will be considered such that unless it can be unequivooilly determined that the medication started and ended prior to the first dose of This document and the partial date (s), the more amore amore an arrival date (s), the mean will be classified as concomitant. To facilitate this decision-making process defined in section 3.1.6.1 will be considered.

3.5.2 Withdrawal from study medication will be classified as concomitant. To facilitate this decision-making process

Reasons for premature withdrawal from the study for randomized subjects are collected on the eCRF and include the following fields:

- Subject decision
- Adverse event
- Severe non-compliance to protocol

Other

Randomized subjects who withdraw prior to Visit 3 are asked to complete and early withdrawal TC (see Table 1).

Subjects who withdraw prior to randomization, or are lost to follow-up following Visit 3 (i.e. the safety follow-up call) will have their end of study status collected in the eCRF under the following fields:

Adverse event

Death

Lost to follow-up

Physician decision

Protocol \*\* Subjects who withdraw prior to randomization, or are lost to follow-up following Visit 3 (i.e. the safety follow-up call) will have their end of study status collected in the eCRF under the following fields:

Adverse event

Death

Lost to follow-up

Physician decision

Protocol deviation

Screen failure

Site terminated by species or

- Site terminated by specisor
- Study terminated
- Withdrawal by subject
- Withdraw by parent/guardian
- Non-sompliance with study drug

# Screen Failures

• no mpliant of the specify)

document in the specify of the specify of the specify of the specific of the spe Screen failures are subjects who do not fulfill the eligibility criteria for the study, and therefore must not be randomized. These subjects should be recorded as a 'Screen Failure' on the disposition eCRF page. Subjects who are screen failures may be re-screened once if

temporary reasons for the original screen failure (eg, respiratory infections, asthma exacerbations, episodes of unstable asthma) have resolved.

If a subject is in screening and cannot complete the randomization visit within 14 days due to local COVID-19 lockdown restrictions, the screening period may be extended to a maximum of 6 weeks. In the event of an extension to the screening period >14 days due to COVID-19, laboratory assessments, vital signs, concomitant medications, and medical/surgical history.

Where a subject does not meet all the all

Where a subject does not meet all the eligibility criteria but is randomized in error, or incorrectly started on treatment, the investigator of collections and the investigator of collections. incorrectly started on treatment, the investigator should inform the medical monitor immediately, and a discussion should occur between the medical monitor and the investigator regarding whether to continue or withdraw the subject in the study. The medical monitor must ensure all decisions are appropriately documented. All subjects randomized erroneously will be marked as major PDs, considered as IPDs and will be analyzed in Cordance with the PK and Safety analysis set definitions (Section 2.1).

#### 4. ANALYSIS METHODS

#### 4.1 Statistical Considerations

Analyses described within this Statistical Aralysis Plan will be performed by

The study is descriptive. There are no productived statistical hypotheses and/or decision rules.

4.1.1 Treatment groups

Descriptive summaries and analysis of endpoints listed below will be grouped by treatment. As subjects will receive both ROA MDI 160/180 and Pulmicort Respules, they will be represented by the treatment they receive at each visit. Therefore, post-randomization analyses of endpoints will not be woken down by visits, since visits will be mutually exclusive per subject and their dosed treatment combinations.

Unless stated enerwise, listings will be grouped by randomized treatment sequence and visit.

# Analysis methods

peatment they received. Any subjects who are erroneously randomized will be identified as major PDs, considered as IPDs and listed in the CSR.

Unless otherwise stated, descriptive summaries of continuous endpoints will include: The number of subjects included in the analysis (n); Mean; Standard Deviation; Median; Minimum; Maximum. Summaries of categorical endpoints will include the absolute counts and percentage, with the denominator used in the percentage calculation clearly defined in the footnote of the table. Unless stated otherwise, the denominator will be the number of subjects in the analysis set used for the descriptive summary.

#### 4.2.1 Subject Disposition

an subjects who have been enrolled and have screen failed will be summarized. The number of subjects who were enrolled, screened and screen failed will be summarized. The number and percentage of subjects will be presented by the following categories; randomized, included in PK analysis set, included in Safety analysis set, not randomized who did randomized who did randomized who did not receive study treatment (and reasons), completed, and discontinued the study (and reasons). For categories that are post-randomization, summaries will be further

split by randomized treatment sequence and overall.

All randomized subjects who were discontinued prematurely will be lightly by randomized treatment sequence including date of, and reason for study discontinuation.

A separate listing will display the planned treatment sequence and the actual treatment received for all randomized subjects.

Additionally, subjects in the safety analysis set who wave excluded from the PK analysis set

will be listed and will include the actual treatment equence and reason for exclusion.

Moreover, data excluded from the PK malyes set will be listed separately for all subjects in the PK analysis set, including actual reatment and reason for exclusion.

4.2.2 Demographic and Baseline Characteristics

The following demographics and subject characteristics will be collected at Visit 1 and Re-

Screening visit, if applicable

Ethnicity

- Weight (kg)
- Height (cm)
- BMI (kg/m<sup>2</sup>)

These variables will be summarized by randomized treatment sequence and overall for all randomized subjects. This summary will be re-produced for subjects in the PK analysis set.

Additionally, the variables above, along with randomized treatment sequence and country,

A standard medical, disease, and surgical history will be recorded on the eCRF at Visit 1. The results of the physical examination at Visit 1 and at unscheduled visits, if applicable will documented in medical history for each subject. Any new abnormal medical physical reported as an AE.

General medical history will be categorized into past and current medical history. Current medical history will be defined as a condition that is either classified con-going or ending after the screening Visit 1.

Medical, disease and surgical history data will be listed by subject including randomized treatment sequence, Medical Dictionary for Regulatory Advities (MedDRA) System Organ Partial dates for the above calculations will be handled as per section 3.1.6.

4.2.2.2 Asthma history

Asthma history Class (SOC), MedDRA Preferred Term, start dat Omd op date (or ongoing if applicable) and

4.2.2.2 Asthma history
Asthma history will be listed separately by subject and will include randomized treatment sequence, date of asthma diagnoses, asthma diagnosed by clinician for at least 3 months prior to Visit 1 (Yes, No), any life meatening asthma episodes prior to Visit 1 (Yes, No), upper respiratory infection involving antibiotic treatment which was not resolved within the 14 days prior to Visit 1 (Yes, No) and associated conditions / triggers / allergies.

# Treament Exposure 4.2.3

Treatment coosure and dosing information will be collected on the eCRF and will be listed for all subjects in the safety analysis set, including dosing date/time, treatment, total dose, overdese (Yes, No).

# Protocol deviations

All randomized subjects with protocol deviations will be listed by randomized treatment sequence, date, visit (if applicable) and reported deviation term and will be sorted by major and minor, with an indication on whether or not the deviation was considered important (Yes, No).

A separate listing including only the COVID-19 related PDs will be produced.

#### 4.2.5 Pharmacokinetics (PK)

The complete PK analysis, derivation and presentation of the associated PK parameters will

Plasma concentration and PK parameter summaries will be based on the PK analysis and Individual plasma concentration and pharmacokinetic parameter listings will be based.

4.2.5.1 Analysis of the plant.

A listing of the plant.

4.2.5.1 Analysis of the plasma concentrations

A listing of the actual PK blood sample collection times, and all reportable budesonide concentrations will be provided for all ability. concentrations will be provided for all children in the safety analysis set. Plasma concentrations outside of the quantification range will be presented as NQ (Not Quantifiable). Concentration data will be presented to 3 significant figures as received from the bioanalytical laboratory.

Plasma concentrations of budesonide will be committeed by treatment and nominal timepoints using the following descriptive statistics:

- ations in the analysis n: Number of evaluable obse
- n-: Number of observations below the lower limit of quantification (LLOQ)
- Mean: Arithmetic mean calculated using untransformed data
- SD: Standard Deviation calculated using untransformed data
- gMean: Geometric mean, calculated as exp[m], where m = mean(log-transformed)
- geV%: Geometric Coefficient of Variation, calculated as 100 √ [exp(s^2)-1], where s is the standard deviation of the data on the log scale
- Median: Median calculated using untransformed data
- Min: Minimum value of the untransformed data
- Max: Maximum value of the untransformed data

NQ observations at any timepoint will be handled as per the rules defined in Section 3.1.6.2. Any NQ observations imputed as 0 will be excluded from the calculation of the geometric mean and the geometric coefficient of variation.

As per the PK analysis plan, at least 66% of observations within the quantification range are required at each timepoint for the descriptive statistics to be calculated. Otherwise the statistics will be set as NC (Not Calculable) and only the minimum and maximum will be presented.

Descriptive statistics will be presented to 4 significant figures (sf's) with the exception of the minimum and maximum which will be presented to 3 sf's and gCV to 1 decimal place.

# Analysis of the primary PK endpoints

The primary endpoints; AUC0-t and Cmax (Section 3.2) for budesonide in the compared separately between treatments with an ANOVA model using the natural logarithm of AUC0-t and Cmax as the response and treatment, treatment sequence, perigon and subject within sequence as fixed effects. Please see example SAS® code belows.

```
proc mixed data=maxfall method=REML;
                                                                                                                    by paramed;
class trtan trtsequent aperiod usubjid(trtsequent);
model log aval = trtan trtsequent aperiod usubjid(trtsequent);
LSmeans trtan / CL alpha=0.05; * Treargent Smean estimates with 95% CI;
LSmeans trtan / diff CL alpha=0.1; * LSmeans t
```

geometric means together with 2-sides 5% confidence intervals for each treatment group. Also, geometric mean ratios between test (BDA MDI) and reference (Pulmicort Respules) treatments, along with the associated 90% confidence limits will be calculated from the models. Moreover, the intra bject coefficient variation (CV%) will be calculated as 100 ×  $\sqrt{[\exp(MSE) - 1]}$ , where MSE is the mean squared error from the model.

The primary treatment comparison of BDA MDI versus Pulmicort Respules for the relative exposure of but sonide will be conducted on the PK analysis set. Only subjects with evaluable Romeasures from both treatment arms will be included in the ANOVA.

parameters). Additionally, the primary PK endpoints will be summarized descriptively as per (4.2.5.3, PK

As this study is primarily descriptive in nature, there are no predefined statistical hypotheses and no predetermined tests or decision rules for the aforementioned analyses.

#### 4.2.5.3 PK parameters

A listing of the derived PK parameters will be provided for all children in the safety analysis set, including treatment and visit, where: Cmax will be presented to the same number of significant figures (sf's) as received from the bioanalytical laboratory; AUC0-t and AUC0-inf

- gMean: Geometric mean, calculated as exp[m], where mean(log-transformed data)
- data) gCV%: Geometric Coefficient of Variation calculated as  $100 \sqrt{[\exp(s^2)-1]}$ , where s is the standard deviation of the data or
- Median: Median calculated using intransformed data
- Min: Minimum value of the untransformed data

  Max: Maximum value of the untransformed data

Descriptive statistics for subjects in the PK analysis set will be presented to 4 significant figures (sf's) with the exception of the minimum and maximum which will be presented to 3 sf's and the gCV% to decimal point. Only median, minimum and maximum will be reported for tmax and tlast

Calculable) and only the minimum and maximum will be presented.

Analysis of safety variables

The analysis of the As per the PR analysis plan, at least 66% of observations per PK parameter are required for the descriptive statistics to be calculated. Otherwise the statistics will be set as NC (Not

The analysis of the safety variables will be based on the safety analysis set and will be reported using the actual treatment associated with the observed data. All data collected prior to study withdrawal will be included in the analyses. Safety data collected during screening will be listed separately.

#### 4.2.6.1 Adverse events

All AEs will be coded using the most recent version of MedDRA dictionary at the time of database lock.

Treatment emergent AEs (TEAEs) will be listed by actual treatment received, MedDRA terror reported term, study day of start of AE, duration of AE, maximum intensity, seriousness of action taken with IMP, causality and outcome.

Additionally, a key subject information of AE, maximum intensity, seriousness of action taken with IMP, causality and outcome.

Additionally, a key subject information listing of all SAEs during the entire study will be created, including, actual treatment received (if and in the study will be created). created, including, actual treatment received (if applicable), corresponding xint, reported term, preferred term, time from start of treatment to onset of AE (days), time from start of treatment to becoming serious (days), outcome, action taken with IMPand causality. Time references are period specific.

Furthermore, subjects with TEAEs, serious TEAEs, TEAEs, Mat led to death, and TEAEs that led to study withdrawal will be separately listed and summarized by SOC and PT.

aun, and TEAEs that SOC and PT.
so be produced for subjects with any TEAE in any of A high-level descriptive summary will also be the following categories:

- Anv TEAE
- Any TEAE with outcome of
- o Any treatment related
- Any TEAE ading to withdrawal from study

Vital sign variables (Section 3.4.1) will be listed by subject, including actual treatment sequence, visit (repeat/unscheduled assessments inclusive), and date/time of the assessments and clinical significance (Yes, No).

Vital signs variables will be descriptively summarized by actual treatment group and timepoint (pre-dose and post-last DV accesses ) timepoint (pre-dose and post-last PK assessment).

#### 4.2.6.3 Laboratory assessments

The clinical chemistry, hematology, and urinalysis assessments will be listed by actual treatment sequence and visit including repeat/unscheduled measurements. The listings will such application include the following information: test name, date/time of measurement, result, result units, clinical significance (Yes, No) as determined by the Investigator, and an indicator variable relative to the normal ranges (Low, Normal, High).

# Prior and Concomitant medication

The number and percentage of subjects who take allowed concomitant medications, and those who take prohibited concomitant medications during the study, will be presented separately by standardized medication name, within generic class (WHO Drug dictionary text). 🗞 each actual treatment sequence. Similarly, a summary of prior medications will be groduced.

Prior and concomitant medication will be listed separately by subject and will include the following information: actual treatment sequence, reported name, coded preferred term, the route of administration, dose (unit), frequency, start and stop date indication, ongoing status (Yes, No) and therapy reason. Any identified prohibited medication will be clearly indicated in the listings.

Descriptive summaries and listings of prior and concentrate medication will be based on the

safety analysis set.

4.2.7 COVID-19 impacts

Blanc is an on-going trial throughout the coronavirus disease 2019 (COVID-19) outbreak.

Due to the design and short study duration, it is not expected that trial data or the analyses will be greatly impacted by the panderanc. Although, it is important to be able to identify any potential intercurrent events de to COVID-19 and to be able to quantify their impact on the study.

# Premature discontinuation due to COVID-19

If a subject canno continue with procedures and scheduled assessments due to COVID-19 post-randomization, they will be withdrawn from the trial and will be asked to complete the early-withdrawal TC. A separate listing of subjects who prematurely withdraw due to COVID-19 will be provided. The listing will detail the reason for withdrawal and relationship The listing of prendomized analysis set. to COVID-19. The listing of premature withdrawals due to COVID-19 will be based on the all

# Adverse events and serious adverse events due to COVID-19

COVID-19 tests for subjects or caregiver/ parent may be conducted proactively prior to inclusion or site visits at any point throughout the study in accordance with local and national guidance. This will be documented as an unscheduled procedure with a positive result recorded as an AE.

Listings of adverse events linked to COVID-19 will be based on the safety analysis sent of such a content of subjects (across sequences). The such are instingtion and sequences are instingted to the safety analysis sent of such and sequences.

Listings of adverse events linked to COVID-19 will be based on the safety analysis sent of such as a sequence of subjects (across sequences). The sequence of subjects (across sequences). The sequence of subjects (across sequences). The sequence of subjects (across sequences). All subjects with a suspected or confirmed diagnosis of COVID-19 will be listed. The listing

total number of subjects (across sequences). The following frequencies and percentages of subjects in the PK analysis set will be presented:

1. Number of subjects affected by COVID-19 [a]

2. Number of premature withdrawals due to COVID-1900

- Number of subjects with COVID-19 related PDs. 3.
- Number of subjects with COVID-19 relater A
- 5. Number of subjects with COVID-19

meet at least one of the listed criteria in points 2-5. [a] Defined as the number of subjects who

# This document must not be used to support any market (%) (%) FROM PROTOCOL

# BLANC Statistical Analysis Plan V1.0 Final Audit Report And ited to the state of the st Created: By: Status: Transaction ID: "BLANC Statistical Analysis Plan V1.0" History VAILLION